CLINICAL TRIAL: NCT00561470
Title: A Multinational, Randomized, Double-blind Study, Comparing the Efficacy of Aflibercept Once Every 2 Weeks Versus Placebo in Patients With Metastatic Colorectal Cancer (MCRC) Treated With Irinotecan / 5-FU Combination (FOLFIRI) After Failure of an Oxaliplatin Based Regimen
Brief Title: Aflibercept Versus Placebo in Combination With Irinotecan and 5-FU in the Treatment of Patients With Metastatic Colorectal Cancer After Failure of an Oxaliplatin Based Regimen
Acronym: VELOUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry); NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC10262; EudraCT 2007-000820-42
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis
Keywords: colorectal cancer; metastatic; anti-angiogenic; irinotecan; 5-FU; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — aflibercept; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo/FOLFIRI (Placebo Comparator): Participants with Metastatic Colorectal Cancer administered Placebo followed by FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) starting on Day 1 of a 2-week cycle until a treatment discontinuation criterion was met
  Interventions: Drug: Placebo; Drug: FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin)
- Aflibercept/FOLFIRI (Experimental): Participants with Metastatic Colorectal Cancer administered Aflibercept followed by FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) starting on Day 1 of a 2-week cycle until a treatment discontinuation criterion was met
  Interventions: Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®); Drug: FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin)

INTERVENTIONS:
Drug: Placebo — 4 mg/kg of sterile aqueous buffered vehicle (pH 6.0) was administered intra venously (IV) over 1 hour on Day 1, every 2 weeks
  Arms: Placebo/FOLFIRI
Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — 4 mg/kg of Aflibercept was administered IV over 1 hour on Day 1, every 2 weeks.
  Arms: Aflibercept/FOLFIRI
Drug: FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) — The FOLFIRI regimen was initiated immediately after Placebo administration on Day 1
  The FOLFIRI regimen included:
  * 180 mg/m² Irinotecan (Campto®, Camptosar®) IV infusion over 90 minutes and dl leucovorin 400 mg/m² (200 mg/m² for the l-isomer form) IV infusion over 2 hours, followed by:
  * 5-FU 400 mg/m² IV bolus given over 2-4 minutes, followed by:
  * 5-FU 2400 mg/m² continuous IV infusion over 46-hours
  Arms: Placebo/FOLFIRI
Drug: FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) — The FOLFIRI regimen was initiated immediately after Aflibercept administration on Day 1
  The FOLFIRI regimen included:
  * 180 mg/m² Irinotecan (Campto®, Camptosar®) IV infusion over 90 minutes and dl leucovorin 400 mg/m² (200 mg/m² for the l-isomer form) IV infusion over 2 hours, followed by:
  * 5-FU 400 mg/m² IV bolus given over 2-4 minutes, followed by:
  * 5-FU 2400 mg/m² continuous IV infusion over 46-hours
  Arms: Aflibercept/FOLFIRI

SUMMARY:
The main objective of the study was to evaluate the effectiveness of aflibercept (versus placebo) in increasing the overall survival in participants with metastatic colorectal cancer treated with FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) and that have previously failed an oxaliplatin based treatment for metastatic disease.

The secondary objectives were to compare progression-free survival, to evaluate overall response rate, to evaluate the safety profile, to assess immunogenicity of intravenous (IV) aflibercept, and to assess pharmacokinetics of IV aflibercept in both treatment arms.

DETAILED DESCRIPTION:
Participants were

* randomized at baseline (treatment was initiated with 3 days of randomization)
* administered treatment in cycles of 14-days till a study withdrawal criterion was met
* followed up 30 days after discontinuation of treatment, and every 8 weeks until death or end of study.

The criteria for discontinuation of study treatment for a participant are:

* participant (or legal representative) chose to withdraw from treatment
* the investigator thought that continuation of the study would be detrimental to the participants well-being due to

  * disease progression
  * unacceptable AEs
  * intercurrent illnesses
  * non-compliance to the study protocol
* participant was lost to follow-up
* participant was unblinded for the investigational treatment

ELIGIBILITY:
Participants who met the following main selection criteria were included in the study.

Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the colon or rectum
* Metastatic disease that is not amenable to potentially curative treatment
* One and only one prior line of treatment for metastatic disease. This prior line should be an oxaliplatin based chemotherapy (participants who relapse within 6 months of completion of oxaliplatin based adjuvant chemotherapy are eligible)
* Prior treatment with bevacizumab is permitted.

Exclusion Criteria:

* Prior therapy with irinotecan
* Eastern Cooperative Oncology Group performance status >2

The above information is not intended to contain all considerations relevant to participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1226 (Actual)
Dates: Start 2007-11; Primary Completion 2011-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (221):
- United States (87):
  - Sanofi-Aventis Investigational Site Number 840119, Birmingham, Alabama
  - Sanofi-Aventis Investigational Site Number 840074, Muscle Shoals, Alabama
  - Sanofi-Aventis Investigational Site Number 840093, Hot Springs, Arizona
  - Sanofi-Aventis Investigational Site Number 840080, Anaheim, California
  - Sanofi-Aventis Investigational Site Number 840076, Fountain Valley, California
  - Sanofi-Aventis Investigational Site Number 840120, Fountain Valley, California
  - Sanofi-Aventis Investigational Site Number 840073, Greenbrae, California
  - Sanofi-Aventis Investigational Site Number 840101, Hayward, California
  - Sanofi-Aventis Investigational Site Number 840046, La Jolla, California
  - Sanofi-Aventis Investigational Site Number 840116, Loma Linda, California
  - Sanofi-Aventis Investigational Site Number 840048, Long Beach, California
  - Sanofi-Aventis Investigational Site Number 840201, Oakland, California
  - Sanofi-Aventis Investigational Site Number 840901, Roseville, California
  - Sanofi-Aventis Investigational Site Number 840042, Sacramento, California
  - Sanofi-Aventis Investigational Site Number 840301, Sacramento, California
  - Sanofi-Aventis Investigational Site Number 840112, Salinas, California
  - Sanofi-Aventis Investigational Site Number 840006, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840106, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840206, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840306, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840406, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840506, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840606, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840706, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840806, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840906, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840401, San Francisco, California
  - Sanofi-Aventis Investigational Site Number 840601, San Jose, California
  - Sanofi-Aventis Investigational Site Number 840501, Santa Clara, California
  - Sanofi-Aventis Investigational Site Number 840801, South San Francisco, California
  - Sanofi-Aventis Investigational Site Number 840001, Vallejo, California
  - Sanofi-Aventis Investigational Site Number 840701, Walnut Creek, California
  - Sanofi-Aventis Investigational Site Number 840071, Stamford, Connecticut
  - Sanofi-Aventis Investigational Site Number 840014, Newark, Delaware
  - Sanofi-Aventis Investigational Site Number 840089, Boynton Beach, Florida
  - Sanofi-Aventis Investigational Site Number 840041, Gainesville, Florida
  - Sanofi-Aventis Investigational Site Number 840031, Gainesville, Florida
  - Sanofi-Aventis Investigational Site Number 840122, Miami, Florida
  - Sanofi-Aventis Investigational Site Number 840079, The Villages, Florida
  - Sanofi-Aventis Investigational Site Number 840087, Chicago, Illinois
  - Sanofi-Aventis Investigational Site Number 840019, Decatur, Illinois
  - Sanofi-Aventis Investigational Site Number 840115, Elk Grove Village, Illinois
  - Sanofi-Aventis Investigational Site Number 840010, Naperville, Illinois
  - Sanofi-Aventis Investigational Site Number 840113, Quincy, Illinois
  - Sanofi-Aventis Investigational Site Number 840072, Indianapolis, Indiana
  - Sanofi-Aventis Investigational Site Number 840047, Indianapolis, Indiana
  - Sanofi-Aventis Investigational Site Number 840034, Munster, Indiana
  - Sanofi-Aventis Investigational Site Number 840088, Louisville, Kentucky
  - Sanofi-Aventis Investigational Site Number 840096, Paducah, Kentucky
  - Sanofi-Aventis Investigational Site Number 840043, Baton Rouge, Louisiana
  - Sanofi-Aventis Investigational Site Number 840084, Metairie, Louisiana
  - Sanofi-Aventis Investigational Site Number 840015, New Orleans, Louisiana
  - Sanofi-Aventis Investigational Site Number 840070, Rockville, Maryland
  - Sanofi-Aventis Investigational Site Number 840029, Salisbury, Maryland
  - Sanofi-Aventis Investigational Site Number 840053, Pontiac, Michigan
  - Sanofi-Aventis Investigational Site Number 840021, Saint Louis Park, Minnesota
  - Sanofi-Aventis Investigational Site Number 840081, Kansas City, Missouri
  - Sanofi-Aventis Investigational Site Number 840052, St Louis, Missouri
  - Sanofi-Aventis Investigational Site Number 840114, St Louis, Missouri
  - Sanofi-Aventis Investigational Site Number 840049, Las Vegas, Nevada
  - Sanofi-Aventis Investigational Site Number 840044, Albuquerque, New Mexico
  - Sanofi-Aventis Investigational Site Number 840036, Albany, New York
  - Sanofi-Aventis Investigational Site Number 840094, Lake Success, New York
  - Sanofi-Aventis Investigational Site Number 840017, Syracuse, New York
  - Sanofi-Aventis Investigational Site Number 840097, Syracuse, New York
  - Sanofi-Aventis Investigational Site Number 840035, Burlington, North Carolina
  - Sanofi-Aventis Investigational Site Number 840024, Charlotte, North Carolina
  - Sanofi-Aventis Investigational Site Number 840026, Charlotte, North Carolina
  - Sanofi-Aventis Investigational Site Number 840005, Goldsboro, North Carolina
  - Sanofi-Aventis Investigational Site Number 840004, Hendersonville, North Carolina
  - Sanofi-Aventis Investigational Site Number 840075, Winston-Salem, North Carolina
  - Sanofi-Aventis Investigational Site Number 840098, Cincinnati, Ohio
  - Sanofi-Aventis Investigational Site Number 840011, Kettering, Ohio
  - Sanofi-Aventis Investigational Site Number 840086, Middletown, Ohio
  - Sanofi-Aventis Investigational Site Number 840008, Toledo, Ohio
  - Sanofi-Aventis Investigational Site Number 840039, Portland, Oregon
  - Sanofi-Aventis Investigational Site Number 840118, Bethlehem, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840033, Philadelphia, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840012, Pittsburgh, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840082, Pawtucket, Rhode Island
  - Sanofi-Aventis Investigational Site Number 840095, Woonsocket, Rhode Island
  - Sanofi-Aventis Investigational Site Number 840085, Charleston, South Carolina
  - Sanofi-Aventis Investigational Site Number 840037, Spartanburg, South Carolina
  - Sanofi-Aventis Investigational Site Number 840078, Corpus Christi, Texas
  - Sanofi-Aventis Investigational Site Number 840117, Temple, Texas
  - Sanofi-Aventis Investigational Site Number 840099, Seattle, Washington
  - Sanofi-Aventis Investigational Site Number 840002, Marshfield, Wisconsin
- Argentina (4):
  - Sanofi-Aventis Investigational Site Number 032003, Bahía Blanca
  - Sanofi-Aventis Investigational Site Number 032006, Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032005, Ciudad de Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032007, Salta
- Australia (7):
  - Sanofi-Aventis Investigational Site Number 036004, Hornsby
  - Sanofi-Aventis Investigational Site Number 036001, Kingswood
  - Sanofi-Aventis Investigational Site Number 036002, Kurralta Park
  - Sanofi-Aventis Investigational Site Number 036005, Melbourne
  - Sanofi-Aventis Investigational Site Number 036003, Melbourne
  - Sanofi-Aventis Investigational Site Number 036007, Nedlands
  - Sanofi-Aventis Investigational Site Number 036006, Subiaco
- Sanofi-Aventis Investigational Site Number 040001, Vienna, Austria
- Belgium (7):
  - Sanofi-Aventis Investigational Site Number 056006, Bonheiden
  - Sanofi-Aventis Investigational Site Number 056007, Brussels
  - Sanofi-Aventis Investigational Site Number 056002, Brussels
  - Sanofi-Aventis Investigational Site Number 056004, Brussels
  - Sanofi-Aventis Investigational Site Number 056001, Ghent
  - Sanofi-Aventis Investigational Site Number 056005, Haine-Saint-Paul
  - Sanofi-Aventis Investigational Site Number 056003, Leuven
- Brazil (8):
  - Sanofi-Aventis Investigational Site Number 076004, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076005, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076002, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076008, Rio de Janeiro
  - Sanofi-Aventis Investigational Site Number 076003, Rio de Janeiro
  - Sanofi-Aventis Investigational Site Number 076001, Santo André
  - Sanofi-Aventis Investigational Site Number 076007, São Paulo
  - Sanofi-Aventis Investigational Site Number 076006, São Paulo
- Chile (5):
  - Sanofi-Aventis Investigational Site Number 152002, Santiago
  - Sanofi-Aventis Investigational Site Number 152003, Santiago
  - Sanofi-Aventis Investigational Site Number 152001, Santiago
  - Sanofi-Aventis Investigational Site Number 152005, Santiago
  - Sanofi-Aventis Investigational Site Number 152004, Viña del Mar
- Czechia (3):
  - Sanofi-Aventis Investigational Site Number 203002, Brno
  - Sanofi-Aventis Investigational Site Number 203001, Brno
  - Sanofi-Aventis Investigational Site Number 203004, Prague
- Denmark (2):
  - Sanofi-Aventis Investigational Site Number 208003, Aalborg
  - Sanofi-Aventis Investigational Site Number 208001, Odense C
- Estonia (2):
  - Sanofi-Aventis Investigational Site Number 233002, Tallinn
  - Sanofi-Aventis Investigational Site Number 233001, Tartu
- France (5):
  - Sanofi-Aventis Investigational Site Number 250002, Brest
  - Sanofi-Aventis Investigational Site Number 250004, Clichy Cx
  - Sanofi-Aventis Investigational Site Number 250005, La Roche-sur-Yon
  - Sanofi-Aventis Investigational Site Number 250001, Lyon
  - Sanofi-Aventis Investigational Site Number 250003, Paris
- Germany (6):
  - Sanofi-Aventis Investigational Site Number 276003, Aschaffenburg
  - Sanofi-Aventis Investigational Site Number 276002, Essen
  - Sanofi-Aventis Investigational Site Number 276001, Halle
  - Sanofi-Aventis Investigational Site Number 276005, Magdeburg
  - Sanofi-Aventis Investigational Site Number 276004, Magdeburg
  - Sanofi-Aventis Investigational Site Number 276006, München
- Greece (5):
  - Sanofi-Aventis Investigational Site Number 300005, Athens
  - Sanofi-Aventis Investigational Site Number 300004, Athens
  - Sanofi-Aventis Investigational Site Number 300001, Heraklion
  - Sanofi-Aventis Investigational Site Number 300002, Ilion, Athens
  - Sanofi-Aventis Investigational Site Number 300003, Pátrai
- Italy (8):
  - Sanofi-Aventis Investigational Site Number 380007, Ancona
  - Sanofi-Aventis Investigational Site Number 380005, Aviano
  - Sanofi-Aventis Investigational Site Number 380004, Candiolo
  - Sanofi-Aventis Investigational Site Number 380003, Genova
  - Sanofi-Aventis Investigational Site Number 380001, Milan
  - Sanofi-Aventis Investigational Site Number 380002, Milan
  - Sanofi-Aventis Investigational Site Number 380008, Rozzano
  - Sanofi-Aventis Investigational Site Number 380006, San Giovanni Rotondo
- Netherlands (5):
  - Sanofi-Aventis Investigational Site Number 528004, Amsterdam
  - Sanofi-Aventis Investigational Site Number 528001, Blaricum
  - Sanofi-Aventis Investigational Site Number 528005, Breda
  - Sanofi-Aventis Investigational Site Number 528002, Rotterdam
  - Sanofi-Aventis Investigational Site Number 528003, Sittard-Geleen
- New Zealand (2):
  - Sanofi-Aventis Investigational Site Number 554009, Auckland
  - Sanofi-Aventis Investigational Site Number 554010, Christchurch
- Norway (3):
  - Sanofi-Aventis Investigational Site Number 578002, Bergen
  - Sanofi-Aventis Investigational Site Number 578001, Oslo
  - Sanofi-Aventis Investigational Site Number 578003, Stavanger
- Poland (7):
  - Sanofi-Aventis Investigational Site Number 616005, Częstochowa
  - Sanofi-Aventis Investigational Site Number 616004, Elblag
  - Sanofi-Aventis Investigational Site Number 616007, Krakow
  - Sanofi-Aventis Investigational Site Number 616003, Lodz
  - Sanofi-Aventis Investigational Site Number 616002, Poznan
  - Sanofi-Aventis Investigational Site Number 616006, Rybnik
  - Sanofi-Aventis Investigational Site Number 616001, Wroclaw
- Sanofi-Aventis Investigational Site Number 630001, San Juan, Puerto Rico
- Romania (7):
  - Sanofi-Aventis Investigational Site Number 642004, Alba Iulia
  - Sanofi-Aventis Investigational Site Number 642001, Bucharest
  - Sanofi-Aventis Investigational Site Number 642002, Bucharest
  - Sanofi-Aventis Investigational Site Number 642007, Bucharest
  - Sanofi-Aventis Investigational Site Number 642003, Cluj-Napoca
  - Sanofi-Aventis Investigational Site Number 642006, Iași
  - Sanofi-Aventis Investigational Site Number 642005, Suceava
- Russia (6):
  - Sanofi-Aventis Investigational Site Number 643001, Moscow
  - Sanofi-Aventis Investigational Site Number 643006, Moscow
  - Sanofi-Aventis Investigational Site Number 643002, Moscow
  - Sanofi-Aventis Investigational Site Number 643004, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643003, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643007, Saint Petersburg
- South Africa (7):
  - Sanofi-Aventis Investigational Site Number 710004, Cape Town
  - Sanofi-Aventis Investigational Site Number 710005, Durban
  - Sanofi-Aventis Investigational Site Number 710008, Durban
  - Sanofi-Aventis Investigational Site Number 710001, Parktown
  - Sanofi-Aventis Investigational Site Number 710006, Port Elizabeth
  - Sanofi-Aventis Investigational Site Number 710007, Pretoria
  - Sanofi-Aventis Investigational Site Number 710003, Pretoria
- South Korea (5):
  - Sanofi-Aventis Investigational Site Number 410001, Goyang
  - Sanofi-Aventis Investigational Site Number 410003, Seoul
  - Sanofi-Aventis Investigational Site Number 410005, Seoul
  - Sanofi-Aventis Investigational Site Number 410002, Seoul
  - Sanofi-Aventis Investigational Site Number 410004, Seoul
- Spain (6):
  - Sanofi-Aventis Investigational Site Number 724002, Barakaldo
  - Sanofi-Aventis Investigational Site Number 724005, Barcelona
  - Sanofi-Aventis Investigational Site Number 724001, Barcelona
  - Sanofi-Aventis Investigational Site Number 724006, Madrid
  - Sanofi-Aventis Investigational Site Number 724003, Madrid
  - Sanofi-Aventis Investigational Site Number 724007, Reus
- Sweden (3):
  - Sanofi-Aventis Investigational Site Number 752002, Stockholm
  - Sanofi-Aventis Investigational Site Number 752003, Sundsvall
  - Sanofi-Aventis Investigational Site Number 752001, Uppsala
- Turkey (Türkiye) (5):
  - Sanofi-Aventis Investigational Site Number 792005, Adana
  - Sanofi-Aventis Investigational Site Number 792004, Ankara
  - Sanofi-Aventis Investigational Site Number 792001, Ankara
  - Sanofi-Aventis Investigational Site Number 792002, Izmir
  - Sanofi-Aventis Investigational Site Number 792003, Kayseri
- Ukraine (4):
  - Sanofi-Aventis Investigational Site Number 804005, Dnipropetrovsk
  - Sanofi-Aventis Investigational Site Number 804004, Donetsk
  - Sanofi-Aventis Investigational Site Number 804006, Kharkiv
  - Sanofi-Aventis Investigational Site Number 804002, Kharkiv
- United Kingdom (10):
  - Sanofi-Aventis Investigational Site Number 826001, Aberdeen
  - Sanofi-Aventis Investigational Site Number 826010, Bournemouth
  - Sanofi-Aventis Investigational Site Number 826009, Dudley
  - Sanofi-Aventis Investigational Site Number 826008, London
  - Sanofi-Aventis Investigational Site Number 826004, London
  - Sanofi-Aventis Investigational Site Number 826007, London
  - Sanofi-Aventis Investigational Site Number 826011, London
  - Sanofi-Aventis Investigational Site Number 826002, Manchester
  - Sanofi-Aventis Investigational Site Number 826003, Northwood
  - Sanofi-Aventis Investigational Site Number 826005, Sutton

REFERENCES:
- [Derived] Pu T, Peddle AM, Wirapati P, Tsantoulis P, Wu Q, Hong Y, Samuel L, Desai J, Riener M, Saridaki Z, Cunningham D, Tejpar S. Exploratory biomarker analysis of RAS/BRAF somatic mutations and gene expression signatures for predicting treatment effects of aflibercept in the velour trial. NPJ Precis Oncol. 2026 Jan 13. doi: 10.1038/s41698-025-01253-5. Online ahead of print. PMID 41530374
- [Derived] Lu L, Dercle L, Zhao B, Schwartz LH. Deep learning for the prediction of early on-treatment response in metastatic colorectal cancer from serial medical imaging. Nat Commun. 2021 Nov 17;12(1):6654. doi: 10.1038/s41467-021-26990-6. PMID 34789774
- [Derived] Chau I, Fakih M, Garcia-Alfonso P, Linke Z, Ruiz Casado A, Marques EP, Picard P, Celanovic M, Cartwright T. Safety and Effectiveness of Aflibercept + Fluorouracil, Leucovorin, and Irinotecan (FOLFIRI) for the Treatment of Patients with Metastatic Colorectal Cancer (mCRC) in Current Clinical Practice: OZONE Study. Cancers (Basel). 2020 Mar 11;12(3):657. doi: 10.3390/cancers12030657. PMID 32168980
- [Derived] Ruff P, Van Cutsem E, Lakomy R, Prausova J, van Hazel GA, Moiseyenko VM, Soussan-Lazard K, Dochy E, Magherini E, Macarulla T, Papamichael D. Observed benefit and safety of aflibercept in elderly patients with metastatic colorectal cancer: An age-based analysis from the randomized placebo-controlled phase III VELOUR trial. J Geriatr Oncol. 2018 Jan;9(1):32-39. doi: 10.1016/j.jgo.2017.07.010. Epub 2017 Aug 12. PMID 28807738
- [Derived] Stanel SC, Sjoberg J, Salmonson T, Foggi P, Caleno M, Melchiorri D, Gravanis I, Tzogani K, Pignatti F. European Medicines Agency approval summary: Zaltrap for the treatment of patients with oxaliplatin-resistant metastatic colorectal cancer. ESMO Open. 2017 May 2;2(2):e000190. doi: 10.1136/esmoopen-2017-000190. eCollection 2017. PMID 28761750
- [Derived] Van Cutsem E, Joulain F, Hoff PM, Mitchell E, Ruff P, Lakomy R, Prausova J, Moiseyenko VM, van Hazel G, Cunningham D, Arnold D, Schmoll HJ, Ten Tije AJ, McKendrick J, Kroning H, Humblet Y, Gravalos C, Le-Guennec S, Andria M, Dochy E, Vishwanath RL, Macarulla T, Tabernero J. Aflibercept Plus FOLFIRI vs. Placebo Plus FOLFIRI in Second-Line Metastatic Colorectal Cancer: a Post Hoc Analysis of Survival from the Phase III VELOUR Study Subsequent to Exclusion of Patients who had Recurrence During or Within 6 Months of Completing Adjuvant Oxaliplatin-Based Therapy. Target Oncol. 2016 Jun;11(3):383-400. doi: 10.1007/s11523-015-0402-9. PMID 26706237
- [Derived] Tabernero J, Van Cutsem E, Lakomy R, Prausova J, Ruff P, van Hazel GA, Moiseyenko VM, Ferry DR, McKendrick JJ, Soussan-Lazard K, Chevalier S, Allegra CJ. Aflibercept versus placebo in combination with fluorouracil, leucovorin and irinotecan in the treatment of previously treated metastatic colorectal cancer: prespecified subgroup analyses from the VELOUR trial. Eur J Cancer. 2014 Jan;50(2):320-31. doi: 10.1016/j.ejca.2013.09.013. Epub 2013 Oct 16. PMID 24140268
- [Derived] Van Cutsem E, Tabernero J, Lakomy R, Prenen H, Prausova J, Macarulla T, Ruff P, van Hazel GA, Moiseyenko V, Ferry D, McKendrick J, Polikoff J, Tellier A, Castan R, Allegra C. Addition of aflibercept to fluorouracil, leucovorin, and irinotecan improves survival in a phase III randomized trial in patients with metastatic colorectal cancer previously treated with an oxaliplatin-based regimen. J Clin Oncol. 2012 Oct 1;30(28):3499-506. doi: 10.1200/JCO.2012.42.8201. Epub 2012 Sep 4. PMID 22949147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 19 November 2007 and 16 March 2010, 614 participants were randomized to the placebo arm and 612 participants were randomized to the aflibercept arm.
Groups:
- Placebo/FOLFIRI: Participants with Metastatic Colorectal Cancer administered Placebo followed by FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) every two weeks
- Aflibercept/FOLFIRI: Participants with Metastatic Colorectal Cancer administered 4 mg/kg of Aflibercept, followed by FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin) every two weeks
Period: Overall Study
Arm/Group | Placebo/FOLFIRI | Aflibercept/FOLFIRI
Started | 614 | 612
TREATED | 609 | 607
SAFETY POPULATION | 605 (Treated participants excluding 4 who received at least 1 dose of Aflibercept) | 611 (Treated participants including 4 from Placebo/FOLFIRI who received at least 1 dose of Aflibercept)
ONGOING TREATMENT | 11 (Participants continuing treatment on the cutoff date of the final analysis) | 14 (Participants continuing treatment on the cutoff date of the final analysis)
Completed | 0 (Participants met treatment discontinuation criteria or were ongoing treatment on the cutoff date) | 0 (Participants met treatment discontinuation criteria or were ongoing treatment on the cutoff date)
Not Completed | 614 | 612
Not completed — Adverse Event | 74 | 163
Not completed — Disease progression | 437 | 305
Not completed — poor compliance to protocol | 4 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 21 | 20
Not completed — Consent Withdrawn | 2 | 6
Not completed — Subject request | 43 | 77
Not completed — Metastatic surgery | 10 | 12
Not completed — Unauthorized procedure | 3 | 1
Not completed — Randomized but not treated | 5 | 5
Not completed — Missed visit window | 1 | 4
Not completed — Planning surgery | 1 | 1
Not completed — Ongoing Treatment | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Folfiri: Participants with Metastatic Colorectal Cancer administered Placebo and FOLFIRI (Irinotecan, 5- Fluorouracil, and Leucovorin)
- Aflibercept/Folfiri: Participants with Metastatic Colorectal Cancer administered 4 mg/kg of Aflibercept and FOLFIRI (Irinotecan, 5- Fluorouracil, and Leucovorin)
- Total: Total of all reporting groups
Arm/Group | Placebo/Folfiri | Aflibercept/Folfiri | Total
Number analyzed (Participants) | 614 | 612 | 1226
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10.8) | 59.5 (10.5) | 59.8 (10.7)
Age, Customized [Number; unit: participants]
  <65 years | 376 | 407 | 783
  >=65 but <75 years | 199 | 172 | 371
  >=75 years | 39 | 33 | 72
Sex/Gender, Customized [Number; unit: participants]
  Male | 353 | 365 | 718
  Female | 261 | 247 | 508
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 523 | 548 | 1071
  Black | 27 | 16 | 43
  Asian/Oriental | 51 | 35 | 86
  Other | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 4 | 2 | 6
  AUSTRALIA | 42 | 54 | 96
  AUSTRIA | 3 | 4 | 7
  BELGIUM | 37 | 45 | 82
  BRAZIL | 21 | 27 | 48
  CHILE | 31 | 33 | 64
  CZECH REPUBLIC | 30 | 47 | 77
  DENMARK | 9 | 6 | 15
  ESTONIA | 7 | 3 | 10
  FRANCE | 1 | 1 | 2
  GERMANY | 23 | 12 | 35
  GREECE | 9 | 10 | 19
  ITALY | 26 | 23 | 49
  KOREA, REPUBLIC OF | 39 | 26 | 65
  NETHERLANDS | 20 | 14 | 34
  NEW ZEALAND | 13 | 7 | 20
  NORWAY | 14 | 19 | 33
  POLAND | 24 | 32 | 56
  PUERTO RICO | 4 | 2 | 6
  ROMANIA | 16 | 16 | 32
  RUSSIAN FEDERATION | 35 | 40 | 75
  SOUTH AFRICA | 36 | 31 | 67
  SPAIN | 27 | 28 | 55
  SWEDEN | 10 | 4 | 14
  TURKEY | 4 | 2 | 6
  UKRAINE | 11 | 11 | 22
  UNITED KINGDOM | 47 | 52 | 99
  UNITED STATES | 71 | 61 | 132
Eastern Cooperative Oncology Group (ECOG) performance status score [Number; unit: participants] — The ECOG score assesses how the disease affects a participant's daily living abilities. It ranges from 0-5, with 0 being the best and 5 being the worst outcome. "0" reflects a fully active participant, able to carry on all pre-disease performance without restriction. "1" reflects a participant restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. "2" reflects an ambulatory participant, who is up and about more than 50% of waking hours, and capable of all self-care but unable to carry out any work activities.
  participants
    Participants with ECOG Score = 0 | 350 | 349 | 699
    Participants with ECOG Score = 1 | 250 | 250 | 500
    Participants with ECOG Score = 2 | 14 | 13 | 27
Prior Bevacizumab [Number; unit: participants] — Number of participants randomized in the prior bevacizumab stratum as per the interactive voice response system (IVRS).
  participants
    Yes | 187 | 186 | 373
    No | 427 | 426 | 853

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival was the time interval from the date of randomization to the date of death due to any cause. Once disease progression was documented, participants were followed every 2 months for survival status, until death or until the study cutoff date, whichever came first. The final data cutoff date for the analysis of OS was the date when 863 deaths had occurred (07 February 2011).
  OS was estimated using the Kaplan-Meier method, and the Hazard Ratio was estimated using the Cox Proportional Hazard Model.
Time Frame: From the date of the first randomization until the study data cut-off date, 07 February 2011 (approximately three years)
Population: Intent-to-treat population (ITT) - all participants who gave informed consent and were randomized.
Measure: Median (Inter-Quartile Range); unit: months
Units Other Than Participants: Events (Death)
Arm/Group | Placebo/FOLFIRI | Aflibercept/FOLFIRI
Number analyzed (Participants) | 614 | 612
Number analyzed (Events (Death)) | 460 | 403
months | 12.06 [6.83 to 21.03] | 13.50 [7.62 to 25.59]
Statistical Analysis 1: Comparison: Placebo/FOLFIRI vs Aflibercept/FOLFIRI; Test type: Superiority or Other; p = 0.0032, Stratified Log-Rank test — Stratified Log-Rank test p-value. Stratified on ECOG Performance Status and prior Bevacizumab according to IVRS using the Cox Proportional Hazard Model. Significance threshold was set to 0.0466 using the O'Brien-Fleming alpha spending function; Stratified Hazard Ratio = 0.817, 95.34% CI 2-sided [0.713 to 0.937] — Stratified on ECOG Performance Status (0 vs 1 vs 2) and prior Bevacizumab (yes vs no) according to IVRS using the Cox Proportional Hazard Model. Significance threshold was set to 0.0466 using the O'Brien-Fleming alpha spending function

2. Secondary Outcome: Progression-free Survival (PFS) Assessed by Independent Review Committee (IRC)
Description: PFS was the time interval from the date of randomization to the date of progression, or death from any cause if it occurs before tumor progression is documented. To evaluate disease progression, copies of all tumor imaging sets were systematically collected and assessed by the IRC.
  PFS was analyzed using the Kaplan-Meier method, and the Hazard Ratio was estimated using the Cox Proportional Hazard Model.
  The analysis for PFS was performed as planned when 561 deaths (OS events) had occurred.
Time Frame: From the date of the first randomization until the occurrence of 561 OS events, 06 May 2010 (approximately 30 months)
Population: Intent to Treat (ITT) population included all participants who gave informed consent and were randomized.
Measure: Median (Inter-Quartile Range); unit: months
Units Other Than Participants: First PFS Events
Arm/Group | Placebo/FOLFIRI | Aflibercept/FOLFIRI
Number analyzed (Participants) | 614 | 612
Number analyzed (First PFS Events) | 454 | 393
months | 4.67 [2.60 to 9.10] | 6.90 [3.84 to 10.05]
Statistical Analysis 1: Comparison: Placebo/FOLFIRI vs Aflibercept/FOLFIRI; Test type: Superiority or Other; p = 0.00007, Stratified Log-Rank test — Stratified on ECOG Performance Status (0 vs 1 vs 2) and prior Bevacizumab (yes vs no) according to IVRS; Stratified Hazard ratio = 0.758, 99.99% CI 2-sided [0.578 to 0.995] — Stratified on ECOG Performance Status (0 vs 1 vs 2) and prior Bevacizumab (yes vs no) according to IVRS using the Cox Proportional Hazard Model

3. Secondary Outcome: Overall Objective Response Rate (ORR) Based on the Tumor Assessment by the Independent Review Committee (IRC) as Per Response Evaluation Criteria in Solid Tumours (RECIST) Criteria
Description: The overall ORR was the percentage of evaluable participants who achieved complete response [CR] or partial response [PR] according to RECIST criteria version 1.0.
  * CR reflected the disappearance of all tumor lesions (with no new tumors)
  * PR reflected a pre-defined reduction in tumor burden
  Tumors were assessed by the IRC using Computerized Tomography (CT) scans or Magnetic Resonance Imaging (MRI) scans; and an observed response was confirmed by repeated imaging after 4 - 6 weeks.
Time Frame: From the date of the first randomization until the study data cut-off date, 06 May 2010 (approximately 30 months)
Population: The evaluable patient population (EPP) for tumor response included all randomized participants with measurable disease at study entry, as per IRC evaluation, and with at least one valid post-baseline tumor evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo/FOLFIRI | Aflibercept/FOLFIRI
Number analyzed (Participants) | 530 | 531
percentage of participants | 11.1 [8.5 to 13.8] | 19.8 [16.4 to 23.2]
Statistical Analysis 1: Comparison: Placebo/FOLFIRI vs Aflibercept/FOLFIRI; Test type: Superiority or Other; p = 0.0001, Stratified Cochran-Mantel-Haenszel; Stratified on ECOG Performance Status (0 vs 1 vs 2) and Prior Bevacizumab (yes vs no) according to IVRS

4. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: All AEs regardless of seriousness or relationship to study treatment, spanning from the first administration of study treatment until 30 days after the last administration of study treatment, were recorded, and followed until resolution or stabilization.
  The number of participants with all treatment emergent adverse events (TEAE), serious adverse events (SAE), TEAE leading to death, and TEAE leading to permanent treatment discontinuation are reported.
Time Frame: From the date of the first randomization up to 30 days after the treatment discontinuation or until TEAE was resolved or stabilized
Population: The safety population was the subset of the ITT population that took at least one dose of study treatment. Analyses was based on the treatment actually received (any participant who received at least one dose of aflibercept, even when receiving the rest of study treatment with placebo, was counted in the aflibercept treatment arm).
Measure: Number; unit: participants
Arm/Group | Placebo/FOLFIRI | Aflibercept/FOLFIRI
Number analyzed (Participants) | 605 | 611
participants
  Treatment-Emergent Adverse Event (TEAE) | 592 | 606
  Serious TEAE | 198 | 294
  TEAE leading to Death | 29 | 37
  TEAE causing permanent treatment discontinuation | 73 | 164

5. Secondary Outcome: Immunogenicity Assessment: Number of Participants With Positive Sample(s) in the Anti-drug Antibodies (ADA) Assay and in the Neutralizing Anti-drug Antibodies (NAb) Assay
Description: Serum samples for immunogenicity assessment were analyzed using a bridging immunoassay to detect ADA. Positive samples in the ADA assay were further analyzed in the NAb assay using a validated, non-quantitative ligand binding assay.
Time Frame: Baseline, every other treatment cycle, 30 days and 90 days after the last infusion of aflibercept/placebo
Population: Immunogenicity population included all participants who were treated and tested for immunogenicity at least once post-baseline.
Measure: Number; unit: participants
Groups:
- Placebo/FOLFIRI: Participants with Metastatic Colorectal Cancer administered Placebo and FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin)
- Aflibercept/FOLFIRI: Participants with Metastatic Colorectal Cancer administered Aflibercept and FOLFIRI (Irinotecan, 5-Fluorouracil, and Leucovorin)
Arm/Group | Placebo/FOLFIRI | Aflibercept/FOLFIRI
Number analyzed (Participants) | 526 | 521
participants
  At least one positive sample in the ADA assay | 18 | 8
  At least one positive sample in the NAb assay | 2 | 1

ADVERSE EVENTS:
Time Frame: From treatment initiation to 7 February, 2011
Arm/Group | Placebo/FOLFIRI | Aflibercept/FOLFIRI
Serious Adverse Events (participants affected / at risk) | 198/605 | 294/611
Other Adverse Events (participants affected / at risk) | 575/605 | 599/611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/FOLFIRI (N=605) | Aflibercept/FOLFIRI (N=611)
Urinary tract infection (Infections and infestations) | 3 | 8
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 11
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 6 | 5
Bronchitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 5 | 4
Sinusitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 8
Gastroenteritis (Infections and infestations) | 2 | 1
Catheter site infection (Infections and infestations) | 0 | 3
Infection (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 5 | 0
Lung infection (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 3
Perirectal abscess (Infections and infestations) | 0 | 3
Subcutaneous abscess (Infections and infestations) | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Emphysematous cystitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Perinephric abscess (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Viral diarrhoea (Infections and infestations) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign neoplasm of cervix uteri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 3 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 19
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 7 | 24
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Hallucination (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Brachial plexopathy (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 10
Deep vein thrombosis (Vascular disorders) | 7 | 7
Hypotension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 2 | 0
Vena cava thrombosis (Vascular disorders) | 2 | 2
Pelvic venous thrombosis (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 2 | 1
Circulatory collapse (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 19
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 14 | 44
Nausea (Gastrointestinal disorders) | 3 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 8
Vomiting (Gastrointestinal disorders) | 7 | 10
Abdominal pain (Gastrointestinal disorders) | 7 | 12
Constipation (Gastrointestinal disorders) | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 6
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 3
Ascites (Gastrointestinal disorders) | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 11 | 10
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 2
Gingivitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 5 | 4
Colitis (Gastrointestinal disorders) | 1 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 5
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 3
Periodontitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0
Mechanical ileus (Gastrointestinal disorders) | 2 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 2
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal obstruction (Gastrointestinal disorders) | 0 | 1
Rectal stenosis (Gastrointestinal disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 4
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 1 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 3 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 2
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 1
Fatigue (General disorders) | 3 | 2
Asthenia (General disorders) | 4 | 5
Pyrexia (General disorders) | 15 | 10
Oedema peripheral (General disorders) | 3 | 0
Disease progression (General disorders) | 14 | 16
Pain (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 2
Malaise (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 1 | 1
Medical device complication (General disorders) | 0 | 1
Death (General disorders) | 1 | 2
Suprapubic pain (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 3
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/FOLFIRI (N=605) | Aflibercept/FOLFIRI (N=611)
Urinary tract infection (Infections and infestations) | 35 | 51
Neutropenia (Blood and lymphatic system disorders) | 202 | 229
Decreased appetite (Metabolism and nutrition disorders) | 143 | 195
Dehydration (Metabolism and nutrition disorders) | 12 | 33
Insomnia (Psychiatric disorders) | 45 | 47
Headache (Nervous system disorders) | 53 | 136
Dizziness (Nervous system disorders) | 53 | 36
Dysgeusia (Nervous system disorders) | 32 | 42
Neuropathy peripheral (Nervous system disorders) | 30 | 34
Lethargy (Nervous system disorders) | 28 | 33
Hypertension (Vascular disorders) | 65 | 250
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 45 | 168
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 20 | 155
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 67
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 | 69
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 45
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 | 38
Diarrhoea (Gastrointestinal disorders) | 335 | 411
Nausea (Gastrointestinal disorders) | 327 | 322
Stomatitis (Gastrointestinal disorders) | 199 | 304
Vomiting (Gastrointestinal disorders) | 199 | 194
Abdominal pain (Gastrointestinal disorders) | 141 | 158
Constipation (Gastrointestinal disorders) | 146 | 135
Abdominal pain upper (Gastrointestinal disorders) | 46 | 63
Dyspepsia (Gastrointestinal disorders) | 56 | 50
Haemorrhoids (Gastrointestinal disorders) | 13 | 34
Proctalgia (Gastrointestinal disorders) | 11 | 32
Alopecia (Skin and subcutaneous tissue disorders) | 182 | 164
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 26 | 67
Rash (Skin and subcutaneous tissue disorders) | 35 | 41
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 17 | 50
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 33 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 69 | 72
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 31
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 34
Proteinuria (Renal and urinary disorders) | 9 | 63
Fatigue (General disorders) | 234 | 292
Asthenia (General disorders) | 77 | 109
Pyrexia (General disorders) | 73 | 77
Oedema peripheral (General disorders) | 42 | 52
Weight decreased (Investigations) | 87 | 195

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 days for abstracts) in advance of any submission, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed ninety days).